CLINICAL TRIAL: NCT04483401
Title: Developmental Coordination Disorder in Preterm Children: Examining Brain Changes With CO-OP Intervention
Brief Title: Premie DCD Imaging Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jill Zwicker, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H16-00358
Record Dates: First submitted 2019-11-07; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Motor Skills Disorders; Premature Birth
Keywords: DCD; Premature Birth; Neuroimaging; Rehabilitation; Motor Skills
MeSH Terms: conditions — Motor Skills Disorders; Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants are either recruited from the Trajectories Study at their 8-year follow-up visit where the Neonatal Follow-Up Team has determined that the child has DCD and meets inclusion criteria for the study, or participants may contact the research coordinator after seeing a recruitment flyer for this study.
  Both groups will receive occupational therapy once weekly for 10 weeks using the published protocol for the CO-OP approach.
Who Masked: Outcomes Assessor
Masking Description: The occupational therapist assessing the filming of child performing their 3 goals at week 1 and 10 will be blinded to which week the the goals were performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist (No Intervention): Waitlist Participants are first allocated to a waitlist condition. After the first MRI scan, participants "wait" for 12 weeks and have a second MRI scan.
- Treatment arm (Experimental): Upon completion on the waitlist time of 12 weeks, participants then are allocated to the treatment group. Participants are assessed by an independent occupational therapist (before and after intervention) and participate in 10 treatment sessions with a treating occupational therapist. Following the post-treatment assessment, participants have a third MRI scan.
  Interventions: Behavioral: Cognitive Orientation to Occupational Performance (CO-OP)

INTERVENTIONS:
Behavioral: Cognitive Orientation to Occupational Performance (CO-OP) — Intervention: CO-OP is a cognitive approach to solving functional motor problems (Polatajko et al., 2001b). Therapists teach children a global problem solving strategy (Goal-Plan-Do-Check) as a framework for developing specific strategies for overcoming motor problems; these strategies are determined after a dynamic performance analysis by the therapist to determine where the "breakdown" is in performing the task. CO-OP intervention will be administered by occupational therapists who have been trained in the CO-OP approach. Children will be seen once weekly for one hour over 12 weeks at as per published protocol (Polatajko et al., 2001b). Parents or caregivers will be encouraged to attend treatment sessions so that therapists can instruct them how to facilitate strategy use between treatment sessions. Children will select three functional motor goals to be addressed over the course of treatment, rating their performance and satisfaction of these goals pre- and post-intervention.
  Arms: Treatment arm

SUMMARY:
This study will leverage a current longitudinal study of brain development in preterm children. In the Miller/Grunau Trajectories study, preterm children are returning for follow-up at 8-9 years. At this appointment, children undergo MRI and neurodevelopmental testing. Children who are identified with DCD at this appointment will be invited to participate in this intervention study. Participants will have a 2nd MRI 12 weeks after the first scan. They will then receive 12 weekly sessions with an occupational therapist, followed by a third MRI.

Children with DCD who were born very preterm (<32 weeks gestational age) who are not part of the Miller/Grunau study are also eligible to participate.

DETAILED DESCRIPTION:
RATIONALE Developmental coordination disorder (DCD) is one of the most common disorders in children (Wann, 2007), affecting 5-6% of the school-age population; this is > 400,000 children in Canada, or 1-2 children in every classroom (American Psychiatric Association, 2013; Statistics Canada, 2013). Compared with children born at term, preterm children (born 2-4 months early) are 6-8 times more likely to develop DCD (Edwards…Zwicker, 2011). DCD significantly interferes with a child's ability to learn motor skills and to perform everyday activities, such as getting dressed, tying shoelaces, using a knife and fork, printing, playing sports, or riding a bicycle. While it was once believed that children would outgrow this condition, longitudinal research has shown that functional difficulties can persist into adolescence and adulthood (Cantell, Smyth, & Ahonen, 2003; Cousins & Smyth, 2003). Furthermore, secondary psychosocial difficulties often develop, including poor self-esteem, depression, anxiety, problems with peers, loneliness, and decreased participation in physical and social activities (Zwicker, Harris, & Klassen, 2013). Up to half of children with DCD will have co-occurring attention deficit hyperactivity disorder (ADHD) (Kadesjo & Gillberg, 1998). As a chronic health condition, DCD often interferes with an individual's function and quality of life across their lifespan (Cousins & Smyth, 2003; Zwicker et al., 2013)

The cause of DCD is not known, and it is under-recognized, under-diagnosed, and under-treated (Blank et al., 2012). In particular, the investigators do not understand the neural basis of DCD, making it difficult to understand why children with DCD struggle to learn motor skills and to determine how to best intervene to optimize function.

To change the negative trajectory of children with DCD, the investigators need a better understanding of the neural basis of DCD, along with further rehabilitation efforts to improve outcomes. Recently, the investigators and others have conducted small neuroimaging studies to begin to understand brain differences in DCD (Querne et al., 2008; Kashiwagi et al., 2009, Zwicker et al., 2010, 2011, 2012b). These studies, while novel and significant in advancing the field of DCD, are limited by small sample sizes. To further define the neural correlates of DCD, the investigators need to perform larger studies and take advantage of new neuroimaging techniques. To date, no studies have examined neural correlates of DCD in the preterm population, a group that is at particularly high risk for the disorder. In addition, brain imaging studies may determine whether improvements in motor function with current "best practice" rehabilitation intervention are associated with changes in brain structure/function. A greater understanding of the neural basis of DCD may result in earlier diagnosis and early rehabilitation to mediate better brain development.

Currently, the investigators have a study underway that assesses whether rehabilitation intervention and improved outcomes in children with DCD are associated with concurrent brain changes (H14-00397). This proposed research extends this study to determine whether preterm children with DCD show similar brain changes.

SPECIFIC OBJECTIVES AND HYPOTHESES

The proposed study (in conjunction with my current DCD-imaging-intervention study: H14-00397) will allow us to compare brain structure and function in full-term children with DCD and in preterm children with the disorder. While the investigators expect similar neural correlates between the two groups, the investigators hypothesize that the preterm DCD may also show unique brain differences, which may affect their response to rehabilitation. The investigators will address two specific objectives as outlined below:

Objective 1: To characterize structural and functional brain differences in full-term and preterm children with DCD.

Hypothesis: In our current study, the investigators hypothesized that, compared to typically-developing children, children with full-term DCD will show smaller cerebellar volume, differences in microstructural development in motor, sensory and cerebellar pathways, and decreased strength of connectivity in resting, default mode, and motor networks. The investigators expect that preterm children will show similar structural and functional brain differences as full-term children with DCD, but that they may also show mild white matter injury.

Approach: The investigators will use magnetic resonance (MR) imaging and advanced MR techniques to characterize brain structure and function; the investigators will use morphometry to measure cerebral and cerebellar volumes, diffusion tensor imaging (DTI) to assess microstructural development, and functional connectivity MRI to measure connectivity in different brain networks. The investigators will also explore fMRI during a mental rotation task and spectroscopy of the basal ganglia.

Objective 2: To determine if current best-practice rehabilitation intervention induces neuroplastic changes in brain structure/function and positive outcomes in preterm children with DCD.

Hypotheses: Compared to their waitlist scan, the investigators expect that post-treatment scans of preterm children will show: (1) strengthened functional connectivity in resting, default mode, and motor networks; (2) increased integrity of the frontal-cerebellar pathway; (3) increased gray matter volume in the dorsolateral prefrontal, motor and cerebellar cortices; and (4) improved performance and satisfaction ratings of child-chosen functional motor goals. The investigators also expect that there will be a positive association between functional improvements and changes in brain structure/function.

Approach: The investigators will measure brain changes at three time points: once before a waiting period as a baseline scan (conducted as part of the Miller-Grunau Trajectories study at age 8-9 years: C05-0579), once immediately before beginning treatment (12 weeks after the first scan), and once after 12 weeks of intervention. As part of treatment, children will identify three functional motor goals as a target for intervention. The investigators will use the Canadian Occupational Performance Measure (COPM; Law et al., 2005) to measure the child's rating of their performance and satisfaction pre- and post-intervention. To supplement the COPM, the investigators will videotape the child performing each of their motor goals before and after intervention, and an independent occupational therapist will use the Performance Quality Rating Scale (PQRS) to objectively measure performance and change in performance (Miller et al., 2001). As a secondary measure, the investigators will evaluate fine and gross motor skills using the Bruininks-Oseretsky Test of Motor Proficiency-2 (BOT-2: Bruininks & Bruininks, 2005).

ELIGIBILITY:
Our targeted sample size is 15.

Inclusion Criteria:

* children who were born very preterm (≤ 32weeks gestational age)
* 8-12 years of age
* diagnosed with DCD (either in the community or at the Neonatal Follow-Up Program at BC Women's Hospital as part as of the Miller/Grunau Trajectories study)
* live in the Greater Vancouver or surrounding areas

Exclusion Criteria:

* children with other diagnoses that may confound the results (e.g., intellectual disability, visual impairment)
* children who have metal anywhere in their body

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2016-05-26 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 12 weeks
  Children will rate performance and satisfaction (10 point Likert scale) of their three motor goals. The OT calculates an average COPM performance score and satisfaction score. These typically range between 1 and 10, and 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction. A change of 2 points indicates a clinically significant change.
Diffusion Tensor Imaging | 12 weeks
  Fractional anisotrophy and diffusivity (mean, axial and radial)

SECONDARY OUTCOMES:
Bruininks Osteretsky Test of Motor Proficiency (BOT-2) | 12 weeks
  Standardized assessment of motor skills. The investigators will measures fine and gross motor skills using the short form of the BOT-2 which assesses 14 items divided between fine manual control, manual coordination, body coordination, and strength/agility. The results are both Standard Score and Percentile Rank. The higher percentile means better motor skills.
Performance Quality Rating Scale (PQRS) | 12 weeks
  Qualitative observations of movement quality. An independent occupational therapist blinded to the intervention will score the motor performance using the Performance Quality Rating Scale (PQRS) which is composed of Part A, a 10-point performance rating scale to rate actual performance, and Part B, an 11-point magnitude of change scale to rate differences in performance between pre- and post-intervention (down to -5 for worse performance, 0 for no change, and up to +5 for improved performance). A higher change score indicates more improvement. An increase of 3 points is considered clinically significant.
Functional connectivity | 12 weeks
  Spatial independent components analysis of resting state networks
Functional magnetic resonance imaging | 12 weeks
  Patterns of brain activation during mental rotation task
Morphometry (brain volume) | 12 weeks
  White matter, cortical gray matter, deep gray matter, and total volumes for cerebrum and cerebellum

CONTACTS AND LOCATIONS:
Overall Officials: Jill G Zwicker, PhD, OT(C), Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Zwicker JG, Harris SR, Klassen AF. Quality of life domains affected in children with developmental coordination disorder: a systematic review. Child Care Health Dev. 2013 Jul;39(4):562-80. doi: 10.1111/j.1365-2214.2012.01379.x. Epub 2012 Apr 20. PMID 22515477
- [Background] Edwards J, Berube M, Erlandson K, Haug S, Johnstone H, Meagher M, Sarkodee-Adoo S, Zwicker JG. Developmental coordination disorder in school-aged children born very preterm and/or at very low birth weight: a systematic review. J Dev Behav Pediatr. 2011 Nov;32(9):678-87. doi: 10.1097/DBP.0b013e31822a396a. PMID 21900828
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Brain activation of children with developmental coordination disorder is different than peers. Pediatrics. 2010 Sep;126(3):e678-86. doi: 10.1542/peds.2010-0059. Epub 2010 Aug 16. PMID 20713484
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Developmental coordination disorder: a pilot diffusion tensor imaging study. Pediatr Neurol. 2012 Mar;46(3):162-7. doi: 10.1016/j.pediatrneurol.2011.12.007. PMID 22353291
- [Background] Miller LT, Polatajko HJ, Missiuna C, Mandich AD, Macnab JJ. A pilot trial of a cognitive treatment for children with developmental coordination disorder. Hum Mov Sci. 2001 Mar;20(1-2):183-210. doi: 10.1016/s0167-9457(01)00034-3. PMID 11471396
- [Background] Polatajko HJ, Mandich AD, Missiuna C, Miller LT, Macnab JJ, Malloy-Miller T, Kinsella EA. Cognitive orientation to daily occupational performance (CO-OP): part III--the protocol in brief. Phys Occup Ther Pediatr. 2001;20(2-3):107-23. PMID 11345506
- [Background] Wann J. Current approaches to intervention in children with developmental coordination disorder. Dev Med Child Neurol. 2007 Jun;49(6):405. doi: 10.1111/j.1469-8749.2007.00405.x. No abstract available. PMID 17518922
- [Background] Statistics Canada. Population by sex and age group. http://www.statcan.gc.ca/tables-tableaux/sum-som/l01/cst01/demo10a-eng.htm. Published 2014. Accessed January 5, 2015.
- [Background] Cantell MH, Smyth MM, Ahonen TP. Two distinct pathways for developmental coordination disorder: persistence and resolution. Hum Mov Sci. 2003 Nov;22(4-5):413-31. doi: 10.1016/j.humov.2003.09.002. PMID 14624826
- [Background] Cousins M, Smyth MM. Developmental coordination impairments in adulthood. Hum Mov Sci. 2003 Nov;22(4-5):433-59. doi: 10.1016/j.humov.2003.09.003. PMID 14624827
- [Background] Kadesjo B, Gillberg C. Developmental coordination disorder in Swedish 7-year-old children. J Am Acad Child Adolesc Psychiatry. 1999 Jul;38(7):820-8. doi: 10.1097/00004583-199907000-00011. PMID 10405499
- [Background] Blank R, Smits-Engelsman B, Polatajko H, Wilson P; European Academy for Childhood Disability. European Academy for Childhood Disability (EACD): recommendations on the definition, diagnosis and intervention of developmental coordination disorder (long version). Dev Med Child Neurol. 2012 Jan;54(1):54-93. doi: 10.1111/j.1469-8749.2011.04171.x. No abstract available. PMID 22171930
- [Background] Querne L, Berquin P, Vernier-Hauvette MP, Fall S, Deltour L, Meyer ME, de Marco G. Dysfunction of the attentional brain network in children with Developmental Coordination Disorder: a fMRI study. Brain Res. 2008 Dec 9;1244:89-102. doi: 10.1016/j.brainres.2008.07.066. Epub 2008 Jul 29. PMID 18718456
- [Background] Kashiwagi M, Iwaki S, Narumi Y, Tamai H, Suzuki S. Parietal dysfunction in developmental coordination disorder: a functional MRI study. Neuroreport. 2009 Oct 7;20(15):1319-24. doi: 10.1097/WNR.0b013e32832f4d87. PMID 19730138